CLINICAL TRIAL: NCT03022084
Title: Clinical Trial of Sound-Based Versus Behavioral Therapy for Tinnitus
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: VA National Center for Rehabilitative Auditory Research (U.S. Federal Agency)
Collaborators: Desyncra, Inc. (Industry)
Responsible Party: Principal Investigator, Sarah Theodoroff, Research Investigator, VA National Center for Rehabilitative Auditory Research
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PVARF-387005
Record Dates: First submitted 2017-01-12; First posted 2017-01-16 (Estimated); Results first posted 2020-07-13 (Actual); Last update posted 2020-07-13 (Actual); Status verified 2020-06

CONDITIONS: Tinnitus
MeSH Terms: conditions — Tinnitus | interventions — Cognitive Behavioral Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Desyncra (Experimental): This group will use the sound-therapy device, Desyncra™ for Tinnitus Therapy System.
  Interventions: Device: Desyncra
- Cognitive Behavioral Therapy (Other): Standard of Care
  Interventions: Other: Cognitive Behavioral Therapy

INTERVENTIONS:
Device: Desyncra — This group will use the sound-therapy device, Desyncra™ for Tinnitus Therapy System.
  Other Names: Desyncra™ for Tinnitus Therapy System
  Arms: Desyncra
Other: Cognitive Behavioral Therapy — Standard of Care
  Other Names: CBT
  Arms: Cognitive Behavioral Therapy

SUMMARY:
The purpose of this study is to determine if a novel sound-based therapy in comparison to standard of care (cognitive behavioral therapy) results in reducing tinnitus-related effects for people with bothersome tinnitus.

DETAILED DESCRIPTION:
This study is a randomized controlled trial evaluating if a customized sound-therapy device is just as effective or more so, than the standard of care (cognitive behavioral therapy, CBT) for bothersome tinnitus. All eligible participants will be randomly assigned to one of the two groups. Depending on group assignment, participants will attend approximately 7-12 visits over a 7-month period.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years
* Primary and persistent tinnitus (6 months or longer in duration)
* Tonal tinnitus
* Dominant tinnitus frequency measured between 0.2 and 10 kHz
* Tinnitus Questionnaire score
* No current participation in other tinnitus therapy program
* Willing and able to listen to the acoustic prescription for 4-6 hours daily during the trial
* Able to pass the Tone Audibility Assessment with factor of 1.1

Exclusion Criteria:

* Secondary/somatic tinnitus due to a suspected underlying disease
* Atonal, pulsatile, intermittent, or occasional tinnitus
* Any hearing threshold >70 dB HL from .25-8kHz, unless subject passes the Tone Audibility Assessment screening with a factor of 1.1
* Any health or other problems that may prevent the person from completing the study procedures as determined by investigator
* Participant reports current suicidal ideation and/or homicidal ideation
* Use of medication which may trigger tinnitus [e.g., quinine derivatives, aminoglycoside antibiotics, daily high dose non-steroidal anti-inflammatory drugs ≥1000 mg, salicylates (when not prescribed as a low dose for cardiac health), loop diuretics and chemotherapy agents like cis-platin]
* Conductive hearing loss
* Visible congenital or traumatic deformity of the ear
* History of active drainage from the ear within the past 90 days
* History of sudden or rapidly progressive hearing loss within the past 90 days
* Inability to read and respond appropriately to instructions that appear on the computer screen, and/or to perform all of the procedures
* Previous use of Desyncra for Tinnitus Therapy System

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 61 (Actual)
Dates: Start 2017-01; Primary Completion 2019-06 (Actual); Study Completion 2019-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: James Henry (PI), PhD, Principal Investigator — VA RR&D NCRAR; Sarah Theodoroff (Co-PI), PhD, Principal Investigator — VA RR&D NCRAR
Locations (1):
- VA Portland Health Care System, National Center for Rehabilitative Auditory Research, Portland, Oregon, United States

IPD SHARING:
Plan to Share IPD: Undecided

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Desyncra | Cognitive Behavioral Therapy
Started | 29 | 32
Completed | 27 | 29
Not Completed | 2 | 3
Not completed — Lost to Follow-up | 2 | 3

BASELINE CHARACTERISTICS:
Population: Individuals with bothersome tinnitus
Groups:
- Total: Total of all reporting groups
Arm/Group | Desyncra | Cognitive Behavioral Therapy | Total
Number analyzed (Participants) | 29 | 32 | 61
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 22 | 26 | 48
  >=65 years | 7 | 6 | 13
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 13 | 23
  Male | 19 | 19 | 38
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3 | 1 | 4
  Not Hispanic or Latino | 25 | 30 | 55
  Unknown or Not Reported | 1 | 1 | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 1
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 0 | 1
  White | 24 | 29 | 53
  More than one race | 1 | 2 | 3
  Unknown or Not Reported | 2 | 1 | 3
Region of Enrollment [Number; unit: participants]
  United States | 29 | 32 | 61

OUTCOME MEASURES:

1. Primary Outcome: Tinnitus Questionnaire (TQ)
Description: 52-item questionnaire that measures the functional impact of tinnitus (scores range from 0 to 104); lower scores indicate better outcome
Time Frame: 24-weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Desyncra | Cognitive Behavioral Therapy
Number analyzed (Participants) | 27 | 29
score on a scale | 34.3 (16.5) | 35.1 (13.7)
Statistical Analysis 1: Comparison: Desyncra vs Cognitive Behavioral Therapy; Test type: Non-Inferiority — The probability that Desyncra is non-inferior to CBT, defined by the sponsor as the event that mean TQ score change from baseline in the Desyncra arm is no more than 3.5 points worse than the mean TQ change in the CBT arm; Bayesian; Data collected to date were analyzed using a Bayesian approach; Data collected to date were analyzed using a Bayesian approach

ADVERSE EVENTS:
Time Frame: 2 years, 5 months
Arm/Group | Desyncra | Cognitive Behavioral Therapy
All-Cause Mortality (participants affected / at risk) | 0/29 | 0/32
Serious Adverse Events (participants affected / at risk) | 0/29 | 0/32
Other Adverse Events (participants affected / at risk) | 0/29 | 0/32

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-03-13): https://cdn.clinicaltrials.gov/large-docs/84/NCT03022084/Prot_SAP_000.pdf